CLINICAL TRIAL: NCT01516619
Title: Pilot Phase II Trial on Safety and Activity of Secondary Prophylaxis With Romiplostim in Patients With Non-Hodgkin Lymphoma and Chemotherapy-induced Thrombocytopenia
Brief Title: Secondary Prophylaxis in Non-Hodgkin Lymphoma (NHL) and Chemotherapy-induced Thrombocytopenia
Acronym: ProRom
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andres J. M. Ferreri (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Andres J. M. Ferreri, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ProRom
Record Dates: First submitted 2012-01-08; First posted 2012-01-25 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: NHL; chemotherapy-induced grade-4 thrombocytopenia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- romiplostim (Experimental)
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Romiplostim will be administered subcutaneously at a dose of 250 μg on the 1st, 3rd and 5th days after the last day of chemotherapy delivery and, then, every two days until the achievement of 75.000 plt/μL.
  In the case of unsuccessful use of romiplostim after the second chemotherapy course, dose escalation to 500 μg/day, with the same above-mentioned schedule, will be indicated after the third course and for all the further courses, with a maximum of 8.
  Other Names: chemotherapy-induced thrombocytopenia; Nplate

SUMMARY:
This is a monocentric, prospective phase II trial addressing safety and capability to prevent grade-4 Chemotherapy-induced Thrombocytopenia (CIT) of romiplostim in patients with NHL.

DETAILED DESCRIPTION:
High-dose chemotherapy followed by autologous stem cell transplant is considered standard of care for patients with relapsed and/or refractory aggressive lymphomas. High-dose chemotherapy, with or without ASCT, may also be used as upfront chemotherapy according to lymphoma histotype (e.g. primary central nervous system lymphomas, mantle cell lymphomas), advanced stage disease, extranodal involvement, and high IPI. Chemotherapy-induced myelosuppression results in various degrees of neutropenia, anemia, and thrombocytopenia and related complications can lead to hospitalization, impaired quality of life, death, and increased healthcare costs.

While myeloid growth factors have reduced neutropenia and the incidence of neutropenic fever, and erythropoietic agents have reduced anemia and transfusions, chemotherapy-induced thrombocytopenia (CIT) still remains an unmet treatment need.

Thrombocytopenia is significantly associated with increased bleeding risk, platelet transfusions need, chemotherapy dose reductions and treatment delays, which usually compromise therapeutic efficacy. Platelet transfusions are also limited by cost, supply, and associated risks, such as transfusion reactions, transmission of infection, alloimmunization and platelet refractoriness. Alternative strategies are evaluating pharmacologic options to stimulate platelet production and to overcome CIT.

The predominant reason for a low platelet count in cancer patients receiving chemotherapy is a deficiency in platelet production. Megakaryopoiesis, the process of development of mega-karyocytes and production of platelets, involves a highly complex cascade of events, from differentiation of immature progenitors to maturation of megakaryocytes and release of platelets into the bone marrow sinusoids. Cytokines present within specialized bone marrow niches contribute to survival, proliferation, and differentiation of megakaryocytes. In addition to TPO, an essential growth factor for platelet production, there are several other growth factors and cytokines, such as IL-1, IL-3, IL-6, IL-11, and SCF, that contribute towards megakaryopoiesis at different stages of development and maturation. In the last decade, a number of these cytokines have been evaluated for the prevention and treatment of thrombocytopenia. Unfortunately, none has yet provided a commercially available agent with a high therapeutic index.

Despite very promising thrombopoietic activity, the clinical development of first-generation recombinant TPOs was halted due to immunogenicity concerns. This led to the development of TPO agonists with no homology to TPO that can bind the TPO receptors and activate signal-ling, leading to increase in platelet production.

ELIGIBILITY:
Inclusion Criteria:

* Patient with NHL of any histotype, both at diagnosis or at relapse, who experienced grade 4 CIT after the first course of chemotherapy containing high doses of methotrexate, cytarabine, cisplatin, cyclophosphamide and/or ifosfamide, and/or conventional doses of anthracyclines or purine analogs, with or without rituximab. The same type of chemotherapy where the grade 4 CIT occurred will be continued at the same planned doses for a maximum of 8 courses.
* ECOG performance status score </= 3.
* Adequate bone marrow function (ANC >1.000; Hb >9,5 g/dL; PLT > 75.000).

Exclusion Criteria:

* Patients eligible for high-dose chemotherapy, where stem cell support is planned.
* Thrombotic events in the previous 5 years before enrolment.
* Other malignancies diagnosed in the previous 5 years before enrolment.
* Severe concomitant illnesses/medical conditions (e.g. impaired respiratory and/or cardiac function, uncontrolled diabetes mellitus).
* Active infectious disease.
* Impaired liver function (bilirubin >2 x upper normal limit; ALT/AST/GGT > 3 x upper normal limit) at one month from salvage chemotherapy conclusion.
* Impaired renal function (creatinine clearance <50 ml/min) at one month from salvage chemotherapy conclusion.
* Non-cooperative behavior or non-compliance.
* Psychiatric diseases or conditions that might impair the ability to give informed consent.
* Pregnant or lactating females.
* Previous therapy with any TPO-mimetic or similar substances.
* Previous therapy supported by transplant of autologous or allogeneic stem cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
safety | participants will be followed for the duration of experimental treatment, an expected average of 6 months
  evaluation of safety, defined by the incidence of grade >/= 4 adverse events (NCI CTCAE v. 4.02 Dec 2009)

SECONDARY OUTCOMES:
activity | From date of registration until the completion of chemotherapy treatment, an expected average of 6 months
  activity defined by the incidence of grade 4 CIT (</= 25 x 10E9/L) per chemotherapy course during experimental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — San Raffaele Scientific Institute, Milano, Italy
Locations (1):
- Dip. Oncoematologia - Fondazione Centro San Raffaele del Monte Tabor, Milan, Italy